CLINICAL TRIAL: NCT05305846
Title: An Explorative, Single-center, Feasibility Study to Collect Data for the Continuous Development of the Future Bladder Sensor Algorithm in Adults During Urodynamics
Brief Title: Data Collection for Development of a Bladder Sensor During Urodynamics
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Essity Hygiene and Health AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: Neoclassic
Record Dates: First submitted 2022-02-25; First posted 2022-03-31 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-02

CONDITIONS: Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Intervention Model Description: Sample size calculation:
  The sample size (n = 66) has been divided into three subgroups according to BMI: normal weight, overweight and obesity class I and class II; minimum 6 subjects each group.
  Dropouts will be replaced.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TENA-PROTO2 (Experimental): Investigational device. Late prototype
  Interventions: Device: TENA-PROTO2

INTERVENTIONS:
Device: TENA-PROTO2 — During urodynamics, the TENA-PROTO2 will be positioned onto the lower abdomen of patients to collect raw data for the continuous development of the future ultrasound bladder sensor.

SUMMARY:
This is an explorative, single-center, feasibility study using a prototype of a future Bladder Sensor to collect data during urodynamics. Obtained data shall be used for the continuous development of the future Bladder Sensor, which is intended for use for individuals suffering from urinary incontinence.

DETAILED DESCRIPTION:
The purpose of this clinical investigation is to collect raw measurement data of the urinary bladder region of participants (patients who are scheduled for urodynamics and fulfill the in- and exclusion criteria) with the TENA-PROTO2, for the continuous development of an algorithm to determine the bladder filling status with the future Bladder Sensor. Secondarily, safety of the subjects will be continuously documented such as adverse events (AE) and device deficiencies (DD); AEs, Adverse Device Events (ADE), Severe Adverse Events (SAE), Severe Adverse Device effects (SADE), Unanticipated Serious Adverse Device Effects (USADE) and DDs.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who are scheduled for urodynamics
2. Men and women defined by biological sex at birth
3. Individuals at the age of ≥ 18 years
4. BMI >18.5 kg/m² and ≤ 39.9 kg/m²
5. Capability to understand the subject information and to provide conscious informed consent
6. Signed informed consent for study participation and data protection regulations
7. Willingness to conduct a urine pregnancy test for all female subjects <55 years old (Exceptions: the site team determines that the subject is not likely to become pregnant due to e.g., hysterectomy, postmenopausal)
8. Capability and willingness to follow the study protocol and procedure of the urodynamics

Exclusion Criteria:

1. Subjects with breached skin, open wounds, sutures or major scar tissue in the suprapubic region
2. Subjects with suprapubic catheter
3. Subjects with implants that can be affected by electromagnetic interference (e.g. pacemaker)
4. Subjects who are pregnant or breast feeding
5. Known allergies or intolerances to one or several components of the study product
6. Alcohol abuse as reported by subject and/ or suspected by investigator that impacts capability to understand the subject information and to provide conscious informed consent in the discretion of the investigator
7. Drug abuse as reported by subject and/ or suspected by investigator that impacts capability to understand the subject information and to provide conscious informed consent in the discretion of the investigator
8. Objections of the investigator to the subject's participation in the trial due to medical reasons or any other reason for which the subject should not participate in the opinion of the investigator
9. Participation in any clinical investigation with systemic and/or pharmaceutical substances within the last 4 weeks and/or in parallel
10. Sponsors, manufacturers or clinical research organization (CRO) staff

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2024-03-18 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Raw measurement data for the development of an algorithm to determine the bladder filling status | 4 months
  Raw data that has been assessed by the prototype (TENA-PROTO2) will be used to develop a product specific algorithm (R&D outcome) for the future Bladder sensor.

SECONDARY OUTCOMES:
Any adverse event (AE) or device deficiency (DD) | Ongoing documentation after enrolment until end of the measurement day (4 months)
  Documentation of AEs, Adverse Device Events (ADE), Severe Adverse Events (SAE), Severe Adverse Device effects (SADE), Unanticipated Serious Adverse Device Effects (USADE) and DDs. In case on an AE, follow-up will be conducted for 14 days.

CONTACTS AND LOCATIONS:
Overall Officials: Diederick Duijvesz, PhD., Principal Investigator — Canisius Wilhelmina Hospital (CWZ)
Locations (1):
- Canisius Wilhelmina Hospital (CWZ), Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: No